CLINICAL TRIAL: NCT01256840
Title: Caloric Restriction With Optimal Nutrition and Aging Study
Brief Title: Long-term Caloric Restriction and Cellular Aging Markers
Acronym: CRONA
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: UCSF-CHR-10-01323
Record Dates: First submitted 2010-12-02; First posted 2010-12-09 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Calorie Restricting Group
- Normal-eating controls
- Obese comparison group

SUMMARY:
The purpose of this study is to see whether people who have restricted the number of calories they eat for a long period of time, compared to normal-eating and obese people, have markers of cellular aging that look younger.

ELIGIBILITY:
Inclusion Criteria:

* Calorie restricting group: Self-reported caloric restriction for at least two years
* Calorie restriction group: BMI below 23
* Normal eating control: Normal eating (no history of caloric restriction) for two years
* Normal eating control: BMI below 30
* Obese comparison group: BMI above 30
* Obese comparison group: Normal eating (no history of caloric restriction) for two years

Exclusion Criteria:

* Regular smoker for the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample and Calorie Restriction Society
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2010-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Janet Tomiyama, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States

REFERENCES:
- [Background] Incollingo Belsky AC, Epel ES, Tomiyama AJ. Clues to maintaining calorie restriction? Psychosocial profiles of successful long-term restrictors. Appetite. 2014 Aug;79:106-12. doi: 10.1016/j.appet.2014.04.006. Epub 2014 Apr 18. PMID 24747211
- [Background] Tomiyama AJ, Milush JM, Lin J, Flynn JM, Kapahi P, Verdin E, Sinclair E, Melov S, Epel ES. Long-term calorie restriction in humans is not associated with indices of delayed immunologic aging: A descriptive study. Nutr Healthy Aging. 2017 Mar 31;4(2):147-156. doi: 10.3233/NHA-160017. PMID 28447069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Calorie Restriction (CR) participants were recruited from the CR Society International, followers of the CR Way, and by referral from participants.
Pre-assignment Details: Inclusion criteria and indicators for CR were reporting calorie restriction without malnutrition for a minimum of two years, BMI < 24.99, and fasting glucose <80 mg/dL.
Groups:
- Calorie Restricting Group: Inclusion criteria for the CR group were reporting calorie restriction without malnutrition for a minimum of two years and BMI < 24.99. Whenever possible, the President of the CR Way Longevity Center and Vice President for Research of the CR Society International or the Chairman of the Board of The CR Society International and Treasurer and Vice President of the CR Way Longevity Center confirmed each participant's self-reported duration of and adherence to calorie restriction. Calorie restriction was also verified via four weekly random fasting glucose tests (<80 mg/dL) with Bayer glucometers. Nursing staff verified BMI on-site.
- Normal-eating Controls; Obese Comparison Group: We recruited the comparison groups to match the CR group in age, race/ethnicity, gender, and educational attainment. Additionally, we recruited siblings of CR participants to attempt to control for genetic and environmental factors. All participants were non-smokers, and all were not pregnant.
Period: Overall Study
Arm/Group | Calorie Restricting Group | Normal-eating Controls | Obese Comparison Group
Started | 30 | 16 | 25
Completed | 30 | 16 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calorie Restricting Group | Normal-eating Controls | Obese Comparison Group | Total
Number analyzed (Participants) | 30 | 16 | 25 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.64 (15.38) | 49.33 (12.49) | 58.84 (13.98) | 55.01 (14.53)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex information is missing for 2 of the participants - one in the CR group and one in the normal eating group.
  Participants
    number analyzed (Participants) | 29 | 15 | 25 | 69
    Female | 7 | 5 | 3 | 15
    Male | 22 | 10 | 22 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race/Ethnicity data is missing for two participants - one in the CR group and one in the Normal Eating group.
  Participants
    Race: number analyzed (Participants) | 29 | 15 | 25 | 69
    Race: White | 26 | 13 | 24 | 63
    Race: Asian | 3 | 2 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 16 | 25 | 69
  United Kingdom | 1 | 0 | 0 | 1
  Japan | 1 | 0 | 0 | 1
Highest Degree [Count of Participants; unit: Participants]
  High School | 2 | 0 | 1 | 3
  Some college | 2 | 1 | 3 | 6
  Bachelor's | 5 | 6 | 2 | 13
  Master's | 6 | 5 | 2 | 13
  Doctoral | 14 | 2 | 11 | 27
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 19.07 (1.84) | 23.27 (90.21) | 29.03 (3.38) | 23.52 (5.07)
Cytomegalovirus seropositive [Count of Participants; unit: Participants] | 13 | 7 | 13 | 33

OUTCOME MEASURES:

1. Primary Outcome: Telomere Length
Description: This study is not a clinical trial, but the UCSF Committee on Human Research requires registration with clinicaltrials.gov. It is a ONE TIME POINT study, where we get a simple blood draw from people from three groups - calorie restricting, normal eating, and obese. Therefore, there IS NO FOLLOW UP/time frame. The outcome measure is assessed on the day of the study. Telomere length is a marker of cellular aging and is used to understand how the cells are aging. We will investigate whether long-term caloric restriction is associated cross-sectionally with longer telomere length (less aging).
Time Frame: One day
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Calorie Restricting Group | Normal-eating Controls | Obese Comparison Group
Number analyzed (Participants) | 30 | 16 | 25
ratio
  Telomere T/S ratio - peripheral blood mononuclear | 0.96 (0.18) | 1.06 (0.15) | 1.06 (0.23)
  Telomere T/S ratio - granulocyte | 1.22 (0.21) | 1.20 (0.23) | 1.14 (0.22)

ADVERSE EVENTS:
Arm/Group | Calorie Restricting Group | Normal-eating Controls | Obese Comparison Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/16 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/16 | 0/25
Other Adverse Events (participants affected / at risk) | 0/30 | 0/16 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No